CLINICAL TRIAL: NCT02625610
Title: A Phase III Open-label, Multicenter Trial of Maintenance Therapy With Avelumab (MSB0010718C) Versus Continuation of First-line Chemotherapy in Subjects With Unresectable, Locally Advanced or Metastatic, Adenocarcinoma of the Stomach, or of the Gastro-esophageal Junction
Brief Title: Avelumab in First-Line Maintenance Gastric Cancer (JAVELIN Gastric 100)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EMR 100070-007; 2015-003300-23 (EudraCT Number)
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Unresectable, Locally Advanced or Metastatic, Adenocarcinoma of the Stomach, or of the Gastro Esophageal Junction
Keywords: Avelumab; Cancer; Unresectable; Locally advanced; Metastatic; Adenocarcinoma of the stomach; Gastro-esophageal junction
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — avelumab; Oxaliplatin; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + Best Supportive Care (BSC) (Experimental): In Maintenance Phase, participants continued the same regimen of oxaliplatin-fluoropyrimidine doublet chemotherapy (oxaliplatin + 5FU/LV or oxaliplatin + capecitabine) as they received during the Induction Phase until disease progression, significant clinical deterioration, unacceptable toxicity, or discontinuation. Participants who were not deemed eligible to receive chemotherapy at the dose and schedule specified above received BSC alone once every 3 weeks. BSC was defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and was based on Investigator's discretion.
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Capecitabine; Other: Best supportive care
- Avelumab (Experimental): In Maintenance phase, participants received avelumab as a 1-hour intravenous (IV) infusion at 10 milligrams per kilogram (mg/kg) once every 2-week treatment cycle until progressive disease or unacceptable toxicity or discontinuation.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Maintenance Phase: Intravenous (IV) infusion (10 mg/kg over 1 hour) once every 2 weeks.
  Other Names: MSB0010718C; Anti PD-L1
  Arms: Avelumab
Drug: Oxaliplatin — Induction Phase: Oxaliplatin was administered at a dose of 85 mg per square meter (mg/m^2) as a continuous intravenous (IV) infusion on Day 1 along with leucovorin followed by 5-Fluorouracil every 2 weeks up to 12 weeks (or) Oxaliplatin at 130 mg/m^2 IV on Day 1 along with capecitabine twice daily for 2 weeks followed by a 1-week rest period given every 3 weeks up to 12 weeks.
  Maintenance Phase: Participants were continued the same regimen of chemotherapy as they received during the Induction Phase until disease progression, significant clinical deterioration, unacceptable toxicity, or discontinuation.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: 5-Fluorouracil — Induction Phase: 5-Fluorouracil was administered at a dose of 2600 mg/m^2 IV continuous infusion over 24 hours on Day 1 (or) 5-FU at 400 mg/m^2 IV push on Day 1 and 2400 mg/m^2 IV continuous infusion over 46-48 hours (Days 1 and 2) along with oxaliplatin and leucovorin every 2 weeks up to 12 weeks. Maintenance Phase: Participants were continued the same regimen of chemotherapy as they received during the Induction Phase until disease progression, significant clinical deterioration, unacceptable toxicity, or discontinuation.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: Leucovorin — Induction Phase: Leucovorin was administered at a dose of 200 mg/m^2 IV (or) Leucovorin 400 mg/m^2 IV on Day 1 along with oxaliplatin and 5-FU every 2 weeks up to 12 weeks.
  Maintenance Phase: Participants were continued the same regimen of chemotherapy as they received during the Induction Phase until disease progression, significant clinical deterioration, unacceptable toxicity, or discontinuation.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: Capecitabine — Induction Phase: Capecitabine was administered at a dose of 1000 mg/m^2 twice daily for 2 weeks followed by a 1-week rest period given every 3 weeks along with oxaliplatin up to 12 weeks.
  Maintenance Phase: Participants were continued the same regimen of chemotherapy as they received during the Induction Phase every 3 weeks until disease progression, significant clinical deterioration, unacceptable toxicity, or discontinuation.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Other: Best supportive care — Treatment administered with the intent to maximize Quality of Life (QoL) without a specific antineoplastic regimen. These may include for example antibiotics, analgesics, antiemetics, thoracentesis, paracentesis, blood transfusions, nutritional support (including jejunostomy), and focal external-beam radiation for control of pain, cough, dyspnea, or bleeding. Best supportive care were administered per institutional guidelines and participants were visit the clinic every 3 weeks.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: Oxaliplatin — Induction Phase: Oxaliplatin will be administered at a dose of 85 mg per square meter (mg/m^2) as a continuous intravenous (IV) infusion on Day 1 along with leucovorin followed by 5-Fluorouracil every 2 weeks up to 12 weeks (or) Oxaliplatin at 130 mg/m^2 IV on Day 1 along with capecitabine twice daily for 2 weeks followed by a 1-week rest period given every 3 weeks up to 12 weeks.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: 5-Fluorouracil — Induction Phase: 5-Fluorouracil will be administered at a dose of 2600 mg/m^2 IV continuous infusion over 24 hours on Day 1 (or) 5-FU at 400 mg/m^2 IV push on Day 1 and 2400 mg/m^2 IV continuous infusion over 46-48 hours (Days 1 and 2) along with oxaliplatin and leucovorin every 2 weeks up to 12 weeks.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: Leucovorin — Induction Phase: Leucovorin will be administered at a dose of 200 mg/m^2 IV (or) Leucovorin 400 mg/m^2 IV on Day 1 along with oxaliplatin and 5-FU every 2 weeks up to 12 weeks.
  Arms: Chemotherapy + Best Supportive Care (BSC)
Drug: Capecitabine — Induction Phase: Capecitabine will be administered at a dose of 1000 mg/m^2 twice daily for 2 weeks followed by a 1-week rest period given every 3 weeks along with oxaliplatin up to 12 weeks.
  Arms: Chemotherapy + Best Supportive Care (BSC)

SUMMARY:
The purpose of this study was to demonstrate superiority of treatment with avelumab versus continuation of first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants greater than or equal to (>=) 18 years
* Disease must be measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Participants with histologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the stomach or gastro-esophageal junction (GEJ)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry
* Estimated life expectancy of more than 12 weeks
* Adequate haematological, hepatic and renal functions defined by the protocol
* Negative blood pregnancy test at Screening for women of childbearing potential
* Highly effective contraception for both male and female participants if the risk of conception exists
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Prior therapy with any antibody or drug targeting T-cell coregulatory proteins
* Concurrent anticancer treatment or immunosuppressive agents
* Prior chemotherapy for unresectable locally advanced or metastatic adenocarcinoma of the stomach or gastro-esophageal junction (GEJ)
* Tumor shown to be human epidermal growth factor 2 plus (HER2+)
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of enrolment and/or if the participant has not fully recovered from the surgery within 4 weeks of enrolment
* Participants receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the study treatment (with the exception of participants with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to <= 10 mg prednisone daily)
* All participants with brain metastases, except those meeting the following criteria: a. Brain metastases have been treated locally, have not been progressing at least 2 months after completion of therapy, and no steroid maintenance therapy is required, and b. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
* Previous malignant disease (other than gastric cancer) within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder, cervical, colorectal, breast)
* Prior organ transplantation, including allogeneic stem-cell transplantation
* Significant acute or chronic infections
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Persisting toxicity related to prior therapy except alopecia
* Neuropathy Grade > 3
* Pregnancy or lactation
* Known alcohol or drug abuse
* History of uncontrolled intercurrent illness including hypertension, active infection, diabetes
* Clinically significant (i.e., active) cardiovascular disease
* All other significant diseases might impair the participant's tolerance of study treatment
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent and that would limit compliance with study requirements
* Vaccination with live or live/attenuated viruses within 55 days of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
* Legal incapacity or limited legal capacity
* Participants will be excluded from the Induction Phase and the Maintenance Phase if administration of their chemotherapy would be inconsistent with the current local labelling (SmPC) (e.g., in regard to contraindications, warnings/precautions or special provisions) for that chemotherapy. Investigators should check updated labelling via relevant websites at the time of entry into the Induction Phase and the Maintenance Phase
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2015-12-24 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc. a business of Merck KGaA, Darmstadt, Germany
Locations (200):
- United States (35):
  - Comprehensive Blood & Cancer Center, Bakersfield, California
  - Virginia Crosson Cancer Center, Fullerton, California
  - UCLA Medical Center, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - Sansum Clinic, Santa Barbara, California
  - Trio - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Norwalk Hospital, Norwalk, Connecticut
  - UF Health Cancer Center Orlando, Orlando, Florida
  - Memorial West Cancer Institute, Pembroke Pines, Florida
  - University of South Florida - Parent, Tampa, Florida
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Franciscan St. Francis Health Cancer Center, Indianapolis, Indiana
  - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Cotton-O'Neil Clinical Research Center, Hematology and Oncology, Topeka, Kansas
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Mount Sinai - PRIME, Jamaica, New York
  - Clinical Research Alliance, Inc, New York, New York
  - University of Rochester, Rochester, New York
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - TriHealth Hatton Institute, Cincinnati, Ohio
  - Mid Ohio Oncology Hematology, DBA The Mark H. Zangmeister Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Baylor Scott & White Health, Temple, Texas
  - University of Washington - Seattle Cancer Care Alliance, East Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Australia (14):
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Base Hospital, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Monash Medical Centre Clayton, Bentleigh, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Brazil (12):
  - Hospital Infanta Cristina, Badajós, Badajoz
  - NOB - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital São Lucas da PUCRS, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Oncosinos - Clínica de Oncologia - Hospital Regina, Novo Hamburgo, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Câncer de Barretos-Fundação Pio XII, Barretos, São Paulo
  - IMV - Instituto De Medicina Vascular Hospital Mae de Deus, Porto Alegre, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo, São Paulo
- Canada (6):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Royal Victoria Hospital, Barrie, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Cité de la Santé de Laval, Laval, Quebec
  - McGill University - Dept. Oncology Clinical Research Program, Montreal, Quebec
- France (14):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - Hôpital de la Timone, Marseille, Bouches Du Rhone
  - Hôpital Morvan, Brest, Brittany Region
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - CHU Besancon - Hopital Jean Minjoz, Besançon, Doubs
  - CHU Bordeaux, Bordeaux, Gironde
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, Haute Garonne
  - CRLCC Eugene Marquis, Rennes, Ille Et Vilaine
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours, Indre Et Loire
  - ICO - Site René Gauducheau, Angers, Maine Et Loire
  - Hôpital Européen Georges Pompidou, Paris, Paris
  - Hôpital Cochin, Paris, Paris
  - CHU Clermont Ferrand, Clermont-Ferrand, Puy De Dome
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
- Germany (8):
  - Klinikum Esslingen GmbH, Esslingen A. N., Baden-Wurttemberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg
  - Klinikum Bogenhausen, Munich, Bavaria
  - Leopoldina Krankenhaus Schweinfurt, Schweinfurt, Bavaria
  - Krankenhaus Nordwest GmbH, Frankfurt am Main, Hesse
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Marienkrankenhaus Hamburg, Hamburg
- Hungary (8):
  - Pecsi Tudomanyegyetem, Pécs, Baranya
  - Petz Aladar Megyei Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Magyar Honvedseg Egeszsegugyi, Budapest
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (13):
  - Presidio Ospedaliero Garibaldi Nesima, Catania
  - Azienda Socio Sanitaria Territoriale di Cremona (Istituti Ospitalieri di Cremona), Cremona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Seconda Università degli Studi di Napoli, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Ospedale degli Infermi, Rimini
  - Università Campus Bio-Medico di Roma, Roma
  - Azienda Ospedaliera S. Maria Di Terni, Terni
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine
- Japan (15):
  - Chiba Cancer Center, Chiba, Chiba
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Izumi Municipal Hospital, Izumi-shi, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Nat Cancer Ctr Hosp, Chūōku, Tokyo-To
  - Toranomon Hospital, Minatoku, Tokyo-To
  - Kagoshima University Medical And Dental Hospital, Kagoshima
- Romania (11):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca, Cluj
  - S.C Radiotherapy Center Cluj S.R.L, Comuna Floresti, Cluj
  - S.C Centrul de Oncologie Sf. Nectarie S.R.L, Craiova, Dolj
  - Spital Lotus SRL, Ploieşti, Prahova
  - S.C Oncocenter Oncologie Clinica S.R.L, Timișoara, Timiș County
  - S.C Oncomed S.R.L, Timișoara, Timiș County
  - S.C Oncopremium Team S.R.L, Baia Mare
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Hifu Terramed Conformal SRL, Bucharest
  - Institutul Regional de Oncologie Iasi, Iași
- Russia (10):
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg, Leningrado
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg, Leningrado
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - LLC Evimed, Chelyabinsk
  - RBIH "Ivanovo Regional Oncological Dispensary", Ivanovo
  - SBIH " Clinical Oncological Dispensary # 1", Krasnodar
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - SBIH of Stavropol territory "Pyatigorsk Oncological Dispensary", Pyatigorsk
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
- South Korea (12):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Keimyung University Dongsan Hospital, Daegu, Jung-gu
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Medical Center, Daegu
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
- Spain (11):
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO l´Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (8):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Patumwan, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (11):
  - Acibadem Adana Hospital, Adana
  - Adana Numune Training and Research Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Dicle University, Medical faculty, Diyarbakır
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
  - Konya Necmettin Erbakan University Meram Medical Faculty, Konya
  - Inonu Uni. Med. Fac., Malatya
  - Mersin University Medical Faculty, Mersin
- United Kingdom (9):
  - Derriford Hospital, Torquay, Devon
  - Barts Hospital, London, Greater London
  - University College London Hospitals, London, Greater London
  - The Christie, Manchester, Greater Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral, Merseyside
  - Mount Vernon Hospital, Northwood, Middlesex
  - Royal Surrey County Hospital, Guildford, Surrey
  - Ninewells Hospital, Dundee, Tayside Region
  - St James's University Hospital, Leeds, West Yorkshire

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- [Derived] Moehler M, Dvorkin M, Boku N, Ozguroglu M, Ryu MH, Muntean AS, Lonardi S, Nechaeva M, Bragagnoli AC, Coskun HS, Cubillo Gracian A, Takano T, Wong R, Safran H, Vaccaro GM, Wainberg ZA, Silver MR, Xiong H, Hong J, Taieb J, Bang YJ. Phase III Trial of Avelumab Maintenance After First-Line Induction Chemotherapy Versus Continuation of Chemotherapy in Patients With Gastric Cancers: Results From JAVELIN Gastric 100. J Clin Oncol. 2021 Mar 20;39(9):966-977. doi: 10.1200/JCO.20.00892. Epub 2020 Nov 16. PMID 33197226
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR%20100070-007
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 1284 participants were screened for this study. Of which 799 participants received at least 1 dose in the Induction Phase, 499 participants were randomized into maintenance phase of the study.
Groups:
- Chemotherapy + Best Supportive Care (BSC): Oxaliplatin was administered at a dose of 85 mg per square meter (mg/m^2) as a continuous intravenous (IV) infusion on Day 1 along with leucovorin at a dose of 200 mg/m^2 or 400 mg/m^2 on Day 1 followed by 5-Fluorouracil at a dose of 2600 mg/m^2 IV continuous infusion over 24 hours on Day 1 or at 400 mg/m^2 IV push on Day 1 and 2400 mg/m^2 IV continuous infusion over 46-48 hours (Day 1 and 2) every 2 weeks up to 12 weeks (or) Oxaliplatin at 130 mg/m^2 IV on Day 1 along with capecitabine at a dose of 1000 mg/m^2 twice daily for 2 weeks followed by a 1-week rest period given every 3 weeks for up to 12 weeks in Induction phase. In Maintenance Phase, participants continued the same regimen of oxaliplatin-fluoropyrimidine doublet chemotherapy (oxaliplatin + 5FU/Leucovorin (LV) or oxaliplatin + capecitabine) as they received during the Induction Phase until disease progression, significant clinical deterioration, unacceptable toxicity, or discontinuation. Participants who were not deemed eligible to receive chemotherapy at the dose and schedule specified above received BSC alone once every 3 weeks. BSC was defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and was based on Investigator's discretion.
- Avelumab: Oxaliplatin was administered at a dose of 85 mg per square meter (mg/m^2) as a continuous intravenous (IV) infusion on Day 1 along with leucovorin at a dose of 200 mg/m^2 or 400 mg/m^2 on Day 1 followed by 5-Fluorouracil at a dose of 2600 mg/m^2 IV continuous infusion over 24 hours on Day 1 or at 400 mg/m^2 IV push on Day 1 and 2400 mg/m^2 IV continuous infusion over 46-48 hours (Day 1 and 2) every 2 weeks up to 12 weeks (or) Oxaliplatin at 130 mg/m^2 IV on Day 1 along with capecitabine at a dose of 1000 mg/m^2 twice daily for 2 weeks followed by a 1-week rest period given every 3 weeks for up to 12 weeks in Induction phase.
  In Maintenance phase, participants received avelumab as a 1-hour intravenous (IV) infusion at 10 milligrams per kilogram (mg/kg) once every 2-week treatment cycle until progressive disease or unacceptable toxicity or discontinuation.
Period: Overall Study
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Started | 250 | 249
Safety-Maintenance Analysis Set | 238 | 243
Completed | 250 | 249
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants included in treatment arm to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab | Total
Number analyzed (Participants) | 250 | 249 | 499
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (11.70) | 60.7 (11.03) | 60.7 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 168
  Male | 167 | 164 | 331
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 19 | 34
  Not Hispanic or Latino | 213 | 220 | 433
  Unknown or Not Reported | 22 | 10 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 161 | 171 | 332
  Black or African American | 2 | 2 | 4
  Asian | 59 | 61 | 120
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Not collected at this site | 22 | 12 | 34
  Other | 3 | 3 | 6
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from randomization to the date of death due to any cause. For participants who were still alive at the time of data analysis or who were lost to follow-up, OS time was censored at the date of last contact. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: Full analysis set included all randomized participants included in treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 250 | 249
months | 10.9 [9.6 to 12.4] | 10.4 [9.1 to 12.0]
Statistical Analysis 1: Comparison: Chemotherapy + Best Supportive Care (BSC) vs Avelumab; Test type: Superiority; p = 0.1779, Log Rank; The treatment arms were compared using a stratified, 1-sided, log rank Test. The stratification factor was region (Asia versus non Asia); Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.11]

2. Secondary Outcome: Progression Free Survival (PFS) by Independent Review Committee (IRC)
Description: The PFS time was defined as the time from date of randomization until date of the first documentation of progressive disease (PD) or death due to any cause (whichever occurs first). PFS was assessed as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as per IRC. PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: Full analysis set included all randomized participants included in treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 250 | 249
months | 4.4 [4.0 to 5.5] | 3.2 [2.8 to 4.1]
Statistical Analysis 1: Comparison: Chemotherapy + Best Supportive Care (BSC) vs Avelumab; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.85 to 1.28]

3. Secondary Outcome: Best Overall Response (BOR) by Investigator Assessment
Description: BOR was determined by RECIST v1.1 per Investigator assessment and defined as best-confirmed response of any of following: complete response (CR), partial response (PR), stable disease (SD) and PD recorded from date of randomization until disease progression or recurrence. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in SLD of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD is defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or appearance of 1 or more new lesions. PR or CR confirmed at a subsequent tumor assessment, not sooner than 5 weeks after initial documentation or at an assessment later than the next assessment after the initial documentation of PR or CR. SD confirmed at least 6 weeks after randomization. Confirmed PD equal to progression <=2 weeks after date of randomization.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: Full analysis set included all randomized participants included in treatment arm to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 250 | 249
Participants
  Complete response | 5 | 8
  Partial response | 31 | 25
  Stable disease | 117 | 92
  Noncomplete response/non progressive disease | 11 | 10
  Progressive disease | 58 | 85
  Non evaluable | 28 | 29

4. Secondary Outcome: Objective Response Rate (ORR) by Investigator Assessment
Description: The ORR defined as the percentage of all randomized participants with a confirmed best overall response (BOR) of partial response (PR),or complete response (CR) according to RECIST v1.1 and as per Investigator assessment. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: Full analysis set included all randomized participants included in treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 250 | 249
percentage of participants | 14.4 [10.3 to 19.4] | 13.3 [9.3 to 18.1]
Statistical Analysis 1: Comparison: Chemotherapy + Best Supportive Care (BSC) vs Avelumab; Test type: Superiority; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.55 to 1.51]

5. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire Through Composite Index Score up to Safety Follow-up (Up to 152.3 Weeks)
Description: EQ-5D-5L is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive overall composite health state index score, with scores ranging from -0.594 to 1. A higher score indicates better health state.
Time Frame: Baseline, Week 3/4, Week 7, Week 13, Week 19, Week 25, Week 31, Week 37, Week 43, Week 49, Week 55, Week 61, Week 67, End of Treatment ( EOT up to 148 weeks) and Safety Follow-up (Up to 152.3 Weeks)
Population: Health-related quality of life (HRQoL) analysis set included randomized participants who had 1 Maintenance Phase Baseline HRQoL assessment and had at least 1 post-Maintenance Phase Baseline HRQoL questionnaire completed. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 159 | 186
Units on Scale
  Week 3/4 | -0.002 (0.1242) | 0.004 (0.1610)
  Week 7: number analyzed (Participants) | 145 | 157
  Week 7 | -0.032 (0.1644) | -0.009 (0.1588)
  Week 13: number analyzed (Participants) | 89 | 103
  Week 13 | -0.053 (0.1733) | -0.017 (0.1599)
  Week 19: number analyzed (Participants) | 56 | 67
  Week 19 | -0.039 (0.1934) | -0.011 (0.1556)
  Week 25: number analyzed (Participants) | 31 | 61
  Week 25 | -0.049 (0.1797) | 0.014 (0.1518)
  Week 31: number analyzed (Participants) | 26 | 45
  Week 31 | -0.023 (0.1619) | 0.013 (0.1665)
  Week 37: number analyzed (Participants) | 18 | 33
  Week 37 | -0.035 (0.1505) | 0.013 (0.2234)
  Week 43: number analyzed (Participants) | 14 | 30
  Week 43 | -0.046 (0.1360) | 0.058 (0.1990)
  Week 49: number analyzed (Participants) | 11 | 27
  Week 49 | -0.100 (0.1796) | 0.026 (0.1936)
  Week 55: number analyzed (Participants) | 5 | 25
  Week 55 | -0.164 (0.2056) | 0.028 (0.2067)
  Week 61: number analyzed (Participants) | 5 | 21
  Week 61 | -0.091 (0.2229) | 0.031 (0.1364)
  Week 67: number analyzed (Participants) | 6 | 17
  Week 67 | -0.076 (0.2347) | 0.039 (0.1954)
  End Of Treatment: number analyzed (Participants) | 134 | 135
  End Of Treatment | -0.125 (0.2432) | -0.138 (0.2461)
  Safety Follow-Up: number analyzed (Participants) | 70 | 69
  Safety Follow-Up | -0.062 (0.2391) | -0.099 (0.1942)

6. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions Health Outcome Questionnaire Through Visual Analogue Scale up to Safety Follow-up (Up to 152.3 Weeks)
Description: EQ-5D-5L is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 159 | 186
Millimeter
  Week 3/4 | 0.9 (13.94) | 0.6 (13.11)
  Week 7: number analyzed (Participants) | 145 | 157
  Week 7 | -0.5 (13.59) | -2.1 (14.09)
  Week 13: number analyzed (Participants) | 89 | 103
  Week 13 | -3.2 (12.83) | -0.7 (13.41)
  Week 19: number analyzed (Participants) | 56 | 67
  Week 19 | -3.5 (16.39) | -0.1 (14.93)
  Week 25: number analyzed (Participants) | 31 | 61
  Week 25 | -4.5 (15.66) | -1.4 (15.76)
  Week 31: number analyzed (Participants) | 26 | 45
  Week 31 | -2.3 (13.14) | 1.4 (17.61)
  Week 37: number analyzed (Participants) | 18 | 33
  Week 37 | -1.7 (11.78) | 0.9 (20.39)
  Week 43: number analyzed (Participants) | 14 | 30
  Week 43 | -4.4 (11.92) | 3.2 (15.34)
  Week 49: number analyzed (Participants) | 11 | 27
  Week 49 | -2.9 (8.95) | 2.1 (13.04)
  Week 55: number analyzed (Participants) | 5 | 25
  Week 55 | -9.4 (16.32) | 3.4 (16.52)
  Week 61: number analyzed (Participants) | 5 | 21
  Week 61 | -6.4 (18.09) | 3.5 (16.15)
  Week 67: number analyzed (Participants) | 6 | 17
  Week 67 | -7.3 (17.10) | 4.9 (17.31)
  End Of Treatment: number analyzed (Participants) | 135 | 135
  End Of Treatment | -12.2 (22.39) | -10.3 (20.84)
  Safety Follow-Up: number analyzed (Participants) | 70 | 69
  Safety Follow-Up | -8.0 (19.24) | -9.6 (20.30)

7. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status Scale Score up to Safety Follow-up (Up to 152.3 Weeks)
Description: European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnoea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact. The EORTC QLQ-C30 GHS/QoL score ranges from 0 to 100; High score indicates better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 160 | 186
units on a scale
  Week 3/4 | 1.30 (15.486) | 0.85 (15.021)
  Week 7: number analyzed (Participants) | 145 | 157
  Week 7 | -1.44 (14.905) | -1.01 (16.967)
  Week 13: number analyzed (Participants) | 90 | 103
  Week 13 | -2.50 (15.424) | 0.24 (17.637)
  Week 19: number analyzed (Participants) | 57 | 67
  Week 19 | -5.85 (18.363) | 1.37 (18.611)
  Week 25: number analyzed (Participants) | 32 | 61
  Week 25 | -4.43 (15.407) | 0.41 (16.204)
  Week 31: number analyzed (Participants) | 27 | 45
  Week 31 | -3.09 (19.902) | 1.85 (16.938)
  Week 37: number analyzed (Participants) | 18 | 33
  Week 37 | -1.39 (22.186) | 1.77 (19.293)
  Week 43: number analyzed (Participants) | 14 | 30
  Week 43 | -1.19 (12.167) | 3.33 (18.518)
  Week 49: number analyzed (Participants) | 11 | 27
  Week 49 | 1.52 (9.731) | 4.01 (15.907)
  Week 55: number analyzed (Participants) | 5 | 25
  Week 55 | 0.00 (11.785) | 4.00 (15.426)
  Week 61: number analyzed (Participants) | 5 | 21
  Week 61 | -5.00 (13.944) | 2.38 (15.622)
  Week 67: number analyzed (Participants) | 6 | 17
  Week 67 | 0.00 (9.129) | 4.90 (18.413)
  End Of Treatment: number analyzed (Participants) | 135 | 135
  End Of Treatment | -11.54 (23.460) | -11.67 (21.409)
  Safety Follow-Up: number analyzed (Participants) | 71 | 70
  Safety Follow-Up | -7.51 (19.475) | -9.29 (24.881)

8. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Stomach Cancer Specific (EORTC QLQ-STO22 ) Questionnaire Scores up to Safety Follow-up (Up to 152.3 Weeks)
Description: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Stomach Cancer Specific (EORTC QLQ-STO22 ) supplements the EORTC QLQ-C30 to assess symptoms and treatment-related side effects commonly reported in participants. There are 22 questions which comprise 5 scales (dysphagia, pain, reflux symptom, dietary restrictions, and anxiety) and 4 single items (dry mouth, hair loss, taste, body image). Most questions use 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 160 | 186
units on a scale
  Dysphagia: Week 3/4 | 0.76 (13.371) | 0.60 (15.227)
  Dysphagia Week 7: number analyzed (Participants) | 145 | 157
  Dysphagia Week 7 | 2.84 (15.258) | 1.34 (13.453)
  Dysphagia Week 13: number analyzed (Participants) | 90 | 102
  Dysphagia Week 13 | 1.60 (14.090) | 0.65 (12.781)
  Dysphagia Week 19: number analyzed (Participants) | 57 | 66
  Dysphagia Week 19 | -0.58 (15.772) | 1.52 (14.307)
  Dysphagia Week 25: number analyzed (Participants) | 32 | 59
  Dysphagia Week 25 | -1.39 (10.465) | 1.69 (14.852)
  Dysphagia Week 31: number analyzed (Participants) | 27 | 43
  Dysphagia Week 31 | 0.82 (14.755) | 4.39 (20.877)
  Dysphagia Week 37: number analyzed (Participants) | 17 | 33
  Dysphagia Week 37 | -7.19 (17.977) | -0.67 (14.683)
  Dysphagia Week 43: number analyzed (Participants) | 14 | 30
  Dysphagia Week 43 | -4.76 (14.265) | -2.59 (13.270)
  Dysphagia Week 49: number analyzed (Participants) | 11 | 27
  Dysphagia Week 49 | -3.03 (8.736) | 1.23 (13.195)
  Dysphagia Week 55: number analyzed (Participants) | 5 | 25
  Dysphagia Week 55 | 0.00 (13.608) | 0.89 (13.194)
  Dysphagia Week 61: number analyzed (Participants) | 5 | 21
  Dysphagia Week 61 | 0.00 (15.713) | 1.06 (12.123)
  Dysphagia Week 67: number analyzed (Participants) | 6 | 17
  Dysphagia Week 67 | -1.85 (10.924) | 1.31 (17.516)
  Dysphagia End Of Treatment: number analyzed (Participants) | 136 | 134
  Dysphagia End Of Treatment | 7.27 (25.134) | 8.21 (22.633)
  Dysphagia Safety Follow-Up: number analyzed (Participants) | 71 | 69
  Dysphagia Safety Follow-Up | 9.39 (21.467) | 7.25 (19.417)
  Pain Week 3/4 | 1.51 (13.013) | -0.04 (13.465)
  Pain Week 7: number analyzed (Participants) | 145 | 157
  Pain Week 7 | 2.53 (15.351) | 2.60 (15.210)
  Pain Week 13: number analyzed (Participants) | 90 | 102
  Pain Week 13 | 2.96 (14.585) | 0.16 (13.523)
  Pain Week 19: number analyzed (Participants) | 57 | 66
  Pain Week 19 | 3.22 (14.152) | -0.51 (14.088)
  Pain Week 25: number analyzed (Participants) | 32 | 59
  Pain Week 25 | -1.56 (13.789) | -1.55 (17.540)
  Pain Week 31: number analyzed (Participants) | 27 | 43
  Pain Week 31 | 4.01 (19.111) | 0.97 (18.564)
  Pain Week 37: number analyzed (Participants) | 17 | 33
  Pain Week 37 | -4.90 (19.777) | -1.26 (12.346)
  Pain Week 43: number analyzed (Participants) | 14 | 30
  Pain Week 43 | 1.79 (18.251) | -1.94 (14.129)
  Pain Week 49: number analyzed (Participants) | 11 | 27
  Pain Week 49 | 1.52 (5.025) | -0.62 (12.853)
  Pain Week 55: number analyzed (Participants) | 5 | 25
  Pain Week 55 | 0.00 (19.543) | -1.00 (10.012)
  Pain Week 61: number analyzed (Participants) | 5 | 21
  Pain Week 61 | 3.33 (9.501) | -1.59 (13.596)
  Pain Week 67: number analyzed (Participants) | 6 | 17
  Pain Week 67 | 0.00 (12.910) | -0.49 (15.721)
  Pain End Of Treatment: number analyzed (Participants) | 136 | 134
  Pain End Of Treatment | 9.25 (20.853) | 9.45 (22.960)
  Pain Safety Follow-Up: number analyzed (Participants) | 71 | 69
  Pain Safety Follow-Up | 8.22 (18.011) | 10.99 (20.931)
  Reflux Week 3/4 | 1.04 (14.197) | 0.12 (13.571)
  Reflux Week 7: number analyzed (Participants) | 145 | 157
  Reflux Week 7 | 0.31 (14.695) | 0.50 (17.807)
  Reflux Week 13: number analyzed (Participants) | 90 | 102
  Reflux Week 13 | 0.99 (14.098) | -1.09 (15.753)
  Reflux Week 19: number analyzed (Participants) | 57 | 66
  Reflux Week 19 | 1.75 (17.032) | -1.68 (15.377)
  Reflux Week 25: number analyzed (Participants) | 32 | 59
  Reflux Week 25 | 0.69 (14.648) | 1.69 (19.770)
  Reflux Week 31: number analyzed (Participants) | 27 | 43
  Reflux Week 31 | -2.06 (14.791) | -1.29 (18.339)
  Reflux Week 37: number analyzed (Participants) | 17 | 37
  Reflux Week 37 | -6.54 (18.864) | -4.38 (17.773)
  Reflux Week 43: number analyzed (Participants) | 14 | 30
  Reflux Week 43 | -3.17 (15.364) | -5.56 (16.699)
  Reflux Week 49: number analyzed (Participants) | 11 | 27
  Reflux Week 49 | 1.01 (9.236) | -2.06 (16.317)
  Reflux Week 55: number analyzed (Participants) | 5 | 25
  Reflux Week 55 | 2.22 (4.969) | -3.56 (19.699)
  Reflux Week 61: number analyzed (Participants) | 5 | 21
  Reflux Week 61 | 6.67 (9.938) | -6.35 (12.944)
  Reflux Week 67: number analyzed (Participants) | 6 | 17
  Reflux Week 67 | 7.41 (13.456) | 0.00 (19.245)
  Reflux End of Treatment: number analyzed (Participants) | 136 | 134
  Reflux End of Treatment | 3.43 (19.529) | 4.73 (20.455)
  Reflux Safety Follow-up: number analyzed (Participants) | 71 | 69
  Reflux Safety Follow-up | 1.56 (20.254) | 2.90 (19.212)
  Eating Restrictions Week 3/4 | 0.73 (16.279) | 0.13 (15.438)
  Eating Restrictions Week 7: number analyzed (Participants) | 145 | 157
  Eating Restrictions Week 7 | 0.98 (16.123) | -0.27 (15.516)
  Eating Restrictions Week 13: number analyzed (Participants) | 90 | 102
  Eating Restrictions Week 13 | 1.02 (14.234) | 0.00 (14.023)
  Eating Restrictions Week 19: number analyzed (Participants) | 57 | 66
  Eating Restrictions Week 19 | -2.34 (16.648) | -0.63 (11.993)
  Eating Restrictions Week 25: number analyzed (Participants) | 32 | 59
  Eating Restrictions Week 25 | -2.08 (18.208) | -1.55 (15.434)
  Eating Restrictions Week 31: number analyzed (Participants) | 27 | 43
  Eating Restrictions Week 31 | -2.47 (15.814) | 0.39 (14.880)
  Eating Restrictions Week 37: number analyzed (Participants) | 17 | 33
  Eating Restrictions Week 37 | -8.82 (21.943) | -3.28 (15.014)
  Eating Restrictions Week 43: number analyzed (Participants) | 14 | 30
  Eating Restrictions Week 43 | -4.76 (18.115) | -3.89 (13.443)
  Eating Restrictions Week 49: number analyzed (Participants) | 11 | 27
  Eating Restrictions Week 49 | 0.76 (11.459) | -5.25 (12.043)
  Eating Restrictions Week 55: number analyzed (Participants) | 5 | 25
  Eating Restrictions Week 55 | 3.33 (15.138) | -6.00 (12.620)
  Eating Restrictions Week 61: number analyzed (Participants) | 5 | 21
  Eating Restrictions Week 61 | 0.00 (15.590) | -5.56 (12.999)
  Eating Restrictions Week 67: number analyzed (Participants) | 6 | 17
  Eating Restrictions Week 67 | 1.39 (13.351) | -2.45 (19.712)
  Eating Restrictions EOT: number analyzed (Participants) | 136 | 134
  Eating Restrictions EOT | 8.27 (20.898) | 10.01 (22.055)
  Eating Restrictions Safety Follow-up: number analyzed (Participants) | 71 | 69
  Eating Restrictions Safety Follow-up | 7.04 (24.055) | 11.59 (25.050)
  Anxiety Week 3/4 | -0.28 (16.150) | -4.06 (18.030)
  Anxiety Week 7: number analyzed (Participants) | 145 | 157
  Anxiety Week 7 | -1.30 (16.947) | -1.20 (20.580)
  Anxiety Week 13: number analyzed (Participants) | 90 | 102
  Anxiety Week 13 | -0.86 (20.685) | -2.83 (16.300)
  Anxiety Week 19: number analyzed (Participants) | 57 | 66
  Anxiety Week 19 | -1.56 (21.561) | -1.68 (19.220)
  Anxiety Week 25: number analyzed (Participants) | 32 | 59
  Anxiety Week 25 | -2.78 (23.780) | -1.69 (14.562)
  Anxiety Week 31: number analyzed (Participants) | 27 | 43
  Anxiety Week 31 | 4.12 (23.700) | -0.52 (24.119)
  Anxiety Week 37: number analyzed (Participants) | 17 | 33
  Anxiety Week 37 | -3.92 (20.765) | -1.01 (27.409)
  Anxiety Week 43: number analyzed (Participants) | 14 | 30
  Anxiety Week 43 | -3.97 (22.480) | -1.11 (24.474)
  Anxiety Week 49: number analyzed (Participants) | 5 | 25
  Anxiety Week 49 | 0.00 (12.172) | -6.17 (17.792)
  Anxiety Week 55: number analyzed (Participants) | 5 | 25
  Anxiety Week 55 | 2.22 (9.296) | -4.00 (20.000)
  Anxiety Week 61: number analyzed (Participants) | 5 | 21
  Anxiety Week 61 | -4.44 (12.669) | -4.76 (24.488)
  Anxiety Week 67: number analyzed (Participants) | 6 | 17
  Anxiety Week 67 | 9.26 (16.355) | -1.96 (24.918)
  Anxiety End of Treatment: number analyzed (Participants) | 136 | 134
  Anxiety End of Treatment | 4.58 (21.868) | 5.89 (23.939)
  Anxiety Safety Follow-Up: number analyzed (Participants) | 71 | 69
  Anxiety Safety Follow-Up | 5.48 (24.116) | 4.99 (26.234)

9. Secondary Outcome: Maintenance Phase: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in participant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both serious TEAEs and non-serious TEAEs. Number of participants with TEAEs and serious TEAEs were reported.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: Safety-Maintenance Analysis Set included all participants who were administered any dose of the maintenance phase study medication or participants randomized to the chemotherapy arm who are designated to receive BSC only. Participants included in the treatment arm according to study treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 238 | 243
Participants
  Any TEAEs | 214 | 223
  Any Serious TEAE | 75 | 89

10. Secondary Outcome: Maintenance Phase: Number of Participants With Grade Change From Baseline to Worst On-Treatment Grade 4 Hematology Values
Description: Blood samples were collected for the analysis of following hematology parameters: lymphocyte count, neutrophil count, white blood cells, platelet count, lipase, serum amylase, creatinine phosphokinase and creatinine. The hematology parameters were graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case (Grade 4) post Baseline is presented. Only those participants with increase to grade 4 have been presented.
Time Frame: From baseline up to 1276 days
Population: Safety-Maintenance Analysis (SMA) Set included all participants who were administered any dose of the maintenance phase study medication or participants randomized to the chemotherapy arm who are designated to receive BSC only. Participants included in the treatment arm according to study treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 238 | 243
Participants
  lymphocyte count decreased | 0 | 1
  neutrophil count decreased | 6 | 1
  white blood cells decreased | 2 | 0
  platelet count decreased | 1 | 0
  lipase increased | 6 | 8
  serum amylase increased | 3 | 2
  creatinine phosphokinase increased | 0 | 2
  creatinine increased | 0 | 1

11. Secondary Outcome: Maintenance Phase: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs
Description: Vital signs assessment included Systolic blood pressure (SBP), Diastolic blood pressure (DBP) and Pulse Rate (PR). Number of Participants with any potentially clinically significant abnormalities in vital signs were reported. Clinical significance was determined by the investigator.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 238 | 243
Participants
  Increased in Systolic blood pressure | 57 | 62
  Decreased in Systolic blood pressure | 43 | 69
  Increased in Diastolic blood pressure: number analyzed (Participants) | 238 | 242
  Increased in Diastolic blood pressure | 14 | 24
  Decreased in Diastolic blood pressure | 21 | 26
  Increased in pulse rate | 46 | 48
  Decreased in pulse rate | 32 | 30

12. Secondary Outcome: Maintenance Phase: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: ECG parameters included heart rate, pulse rate intervals, QRS interval, QT interval corrected based on Fridericia's formula (QTcF) intervals and QTcB intervals. Clinical significance was determined by the investigator. Number of participants with potentially clinically significant ECG abnormalities were reported.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 238 | 243
Participants
  Decreased heart rate | 0 | 1
  Increased heart rate | 2 | 2
  Increased Pulse Rate interval | 1 | 3
  Increased QRS interval | 5 | 8
  QTcF interval greater than (>)450milisecond (ms)less than or equal to(<=)480ms | 9 | 9
  QTcF interval: > 480 ms <= 500 ms | 2 | 3
  QTcF interval: > 500 ms | 3 | 1
  QTcB Interval: > 450 msec <= 480 msec | 19 | 18
  QTcB Interval: > 480 msec <= 500 msec | 2 | 2
  QTcB Interval: > 500 msec | 5 | 3

13. Secondary Outcome: Maintenance Phase: Number of Participants With Shift in Eastern Cooperative Oncology Group (ECOG) Performance Status Score to 1 or Higher Than 1
Description: ECOG PS score is widely used by doctors and researchers to assess how a participants' disease is progressing, and is used to assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. The score ranges from Grade 0 to Grade 5, where Grade 0 = Fully active, able to carry on all pre-disease performance without restriction, Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (like light house work, office work), Grade 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, Grade 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours and Grade 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair, Grade 5 = Death. Number of participants with shift in ECOG PS Score to 1 or Higher Than 1 were reported.
Time Frame: From randomization into maintenance phase up to 1276 days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
Number analyzed (Participants) | 238 | 243
Participants | 140 | 144

ADVERSE EVENTS:
Time Frame: From randomization into maintenance phase up to 1276 days
Description: Safety-Maintenance Analysis Set included all participants who were administered any dose of the maintenance phase study medication or participants randomized to the chemotherapy arm who are designated to receive BSC only. Participants included in the treatment arm according to study treatment actually received.
Arm/Group | Chemotherapy + Best Supportive Care (BSC) | Avelumab
All-Cause Mortality (participants affected / at risk) | 13/238 | 16/243
Serious Adverse Events (participants affected / at risk) | 75/238 | 89/243
Other Adverse Events (participants affected / at risk) | 203/238 | 191/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Best Supportive Care (BSC) (N=238) | Avelumab (N=243)
Dysphagia (Gastrointestinal disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4
Ascites (Gastrointestinal disorders) | 3 | 3
Colitis (Gastrointestinal disorders) | 0 | 3
Ileus (Gastrointestinal disorders) | 0 | 3
Obstruction gastric (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Gastric stenosis (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Disease progression (General disorders) | 6 | 14
Pyrexia (General disorders) | 2 | 4
Asthenia (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Chemical burn of respiratory tract (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Embolism (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Contrast media reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 3 | 1
Headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Nephrostomy (Surgical and medical procedures) | 0 | 1
Device occlusion (Product Issues) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Best Supportive Care (BSC) (N=238) | Avelumab (N=243)
Nausea (Gastrointestinal disorders) | 52 | 41
Abdominal Pain (Gastrointestinal disorders) | 24 | 34
Vomiting (Gastrointestinal disorders) | 27 | 30
Constipation (Gastrointestinal disorders) | 18 | 28
Diarrhoea (Gastrointestinal disorders) | 39 | 27
Abdominal pain upper (Gastrointestinal disorders) | 5 | 22
Dyspepsia (Gastrointestinal disorders) | 15 | 11
Fatigue (General disorders) | 29 | 35
Asthenia (General disorders) | 24 | 30
Pyrexia (General disorders) | 28 | 28
Chills (General disorders) | 4 | 19
Blood creatine phosphokinase increased (Investigations) | 6 | 19
Gamma-glutamyltransferase increased (Investigations) | 15 | 18
Aspartate aminotransferase increased (Investigations) | 17 | 17
Blood alkaline phosphatase increased (Investigations) | 16 | 17
Blood cholesterol increased (Investigations) | 10 | 15
Lipase increased (Investigations) | 22 | 15
Amylase increased (Investigations) | 13 | 14
Alanine aminotransferase increased (Investigations) | 12 | 13
Weight decreased (Investigations) | 19 | 12
Blood bilirubin increased (Investigations) | 13 | 9
Platelet count decreased (Investigations) | 34 | 6
Neutrophil count decreased (Investigations) | 35 | 4
Headache (Nervous system disorders) | 6 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 42 | 14
Dizziness (Nervous system disorders) | 8 | 13
Paraesthesia (Nervous system disorders) | 22 | 11
Neuropathy peripheral (Nervous system disorders) | 32 | 7
Anaemia (Blood and lymphatic system disorders) | 48 | 35
Neutropenia (Blood and lymphatic system disorders) | 36 | 12
Leukopenia (Blood and lymphatic system disorders) | 17 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 34 | 8
Decreased appetite (Metabolism and nutrition disorders) | 42 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 17
Rash (Skin and subcutaneous tissue disorders) | 5 | 15
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 7 | 18
Insomnia (Psychiatric disorders) | 9 | 16
Hypertension (Vascular disorders) | 6 | 14
Upper respiratory tract infection (Infections and infestations) | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02625610/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT02625610/SAP_001.pdf